CLINICAL TRIAL: NCT05451251
Title: Deep Brain Stimulation for Refractory Trigeminal Neuralgia with a Pontine Lesion: a Pilot Study
Brief Title: Deep Brain Stimulation for Refractory Trigeminal Neuralgia with a Pontine Lesion
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-4672
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Trigeminal Neuralgia
Keywords: Multiple sclerosis; Deep brain stimulation; Pontine lesion
MeSH Terms: conditions — Trigeminal Neuralgia; Multiple Sclerosis | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Deep brain stimulation (Experimental): Implantation of deep brain stimulation lead within the pontine lesion
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — Implantation of deep brain stimulation lead within the pontine lesion

SUMMARY:
The aim of this study is to assess the feasibility of deep brain stimulation for refractory trigeminal neuralgia due to a pontine lesion, as is usually seen in the context of multiple sclerosis.

These patients usually have severe intractable facial pain and current medical and surgical options generally fail to achieve long lasting pain relief.

Hoping to improve pain control in this population, the investigators of this trial propose a novel technique consisting of implanting a deep brain stimulation lead within the pontine lesion to modulate the generation of pain signals.

ELIGIBILITY:
Inclusion Criteria:

* Adults of at least 18 years old
* Refractory trigeminal neuralgia : failure of at least 3 drugs and at least two lesioning surgical interventions (radiosurgery, percutaneous rhizotomy, or open rhizotomy).
* Pontine lesion proved by MRI in contact with trigeminal nerve tract

Exclusion Criteria:

* Absolute contraindication to MRI
* Medical contraindication to the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Demonstrating the feasibility of the intervention by assessing protocol completion without deviation | 24 months
  Protocol completion defined by:
  * Lead implantation with success
  * Adjustment of stimulation parameters to minimize adverse effects
  * Minimal follow-up of 6 months after intervention

SECONDARY OUTCOMES:
Lead implantation accuracy | 24 months
  Difference between target and actual lead position
Pain evolution | 24 months
  Evolution of pain severity after the intervention according to the modified Barrow Neurological Institute (mBNI) grading scale.
Facial numbness | 24 months
  Assessed by the Barrow Neurological Institute Facial Numbness Scale and a Quantitative Sensory Testing (QST) protocol.
Complications | 24 months
  Complications arising from the intervention according to the Common Terminology Criteria for Adverse Events (CTCAE) grading scale.
Quality of life progression | 24 months
  Assessed by the Brief Pain Inventory-Facial (BPI-Facial)
Patient acceptability of the procedure | 24 months
  Assessed by a Likert scale with a maximum score of 8. A low score on this scale indicates low acceptability of the surgical procedure, while a high score indicates high acceptability.
Patient global impression of change | 24 months
  Assessed by The Patient Global Impression of Change (PGIC) questionnaire with a maximum score of 18. A low score indicates a low impression of change while a high score indicates a high impression of change.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Open on request.